CLINICAL TRIAL: NCT00530842
Title: Effect of Inhalation of a Free Combination of Tiotropium Once Daily 18 Mcg and Salmeterol Twice Daily 50 Mcg Versus a Fixed Combination of Fluticasone and Salmeterol Twice Daily (500/50 Mcg) on Static Lung Volumes and Exercise Tolerance in COPD Patients (a Randomised, Double-blind, Double Dummy, 16 (2 x 8) Weeks, Crossover Study).
Brief Title: Effect of Tiotropium Plus Salmeterol vs. Fluticasone/Salmeterol on Static Lung Volumes and Exercise Endurance in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Crossover | Purpose: Treatment
Other Study IDs: 205.334
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

INTERVENTIONS:
Drug: Tiotropium plus Salmeterol
Drug: Fluticasone/Salmeterol

SUMMARY:
The primary objective of this study is to demonstrate that treatment with a free combination of tiotropium and salmeterol provides superior improvement in static lung volumes and exercise tolerance compared to a fixed combination of fluticasone and salmeterol in patients with COPD.

The secondary objective includes assessment of safety.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed an Informed Consent Form in accordance with GCP and local legislative requirements prior to participation in the trial, i.e., prior to pre-trial washout of any restricted medications.
2. The patient has a clinical diagnosis of chronic obstructive pulmonary disease (COPD).
3. The patient has relatively stable, moderate to severe airway obstruction.
4. The patient has a pre-bronchodilator forced expiratory volume in the first second (FEV1) less than or equal to 65% of predicted normal determined at Visit 1 using the following predicted equations (R94-1408):

   1. Males Forced expiratory volume in the first second (FEV1) predicted [Litres (L)] = 4.30 x Height [metres] minus 0.029 x Age [years] minus 2.49
   2. Females Forced expiratory volume in the first second (FEV1) predicted [Litres (L)] = 3.95 x Height [metres] minus 0.025 x Age [years] minus 2.60 and a Thoracic Gas Volume (Functional residual volume) ((TGV)(FRC)) bigger than 120% predicted normal at visit 1 (or historical data not older than 6 month)
   3. Males Thoracic Gas Volume (Functional residual volume) ((TGV(FRC)) pred. [Litres (L)] = 2.34 x Height [metres] + 0.009 x Age [years] minus 1.09
   4. Females Thoracic Gas Volume (Functional residual volume) ((TGV(FRC)) pred. [Litres (L)] = 2.24 x Height [metres] + 0.001 x Age [years] minus 1.00
5. The patient is at least 40 years and less than or equal to 75 years old.
6. The patient has a cigarette smoking history of at least 10 pack-years. A pack-year is defined as the equivalent of smoking one pack of cigarettes per day for a year.
7. The patient is able to perform all specified procedures and able to maintain all necessary records during the study period as required in the protocol.
8. The patient is able to inhale the trial medication from the HandiHaler device.
9. The patient is able to inhale the trial medication from the Diskus/Accuhaler device.

Exclusion Criteria:

1. a significant disease other than chronic obstructive pulmonary disease (COPD). (review contraindications for exercise testing),
2. a recent history of myocardial infarction within one year.
3. a recent history of heart failure, pulmonary oedema, or patients with cardiac arrhythmia or any contraindication to exercise described in the CTProtocol within the last 3.
4. daytime supplemental oxygen.
5. a diagnosis of known active tuberculosis.
6. a history of cancer within the last 5 years.
7. a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
8. thoracotomy with pulmonary resection.
9. an upper respiratory tract infection or an exacerbation of chronic obstructive pulmonary disease (COPD)
10. a known hypersensitivity to anticholinergic drug, ß-adrenergic or corticosteroids, lactose or any other component of the inhalation capsule delivery system.
11. a known symptomatic prostatic hypertrophy or bladder neck obstruction.
12. a known moderate or severe renal insufficiency.
13. a known narrow-angle glaucoma.
14. a known untreated hypokalemia.
15. a known untreated thyrotoxicosis.
16. a history of asthma, allergic rhinitis or atopy, or a total blood eosinophil count larger than 600/mm3.
17. treatment with cromolyn sodium or nedocromil sodium
18. treatment with antihistamines or antileukotrienes.
19. treatment with tiotropium for 1 month before Visit 1.
20. treatment with oral corticosteroid medication.
21. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception
22. a history of or active alcohol or drug abuse.
23. an investigational drug within 1 month or 10 half lives
24. a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnoea.
25. participation in a rehabilitation program for chronic obstructive pulmonary disease (COPD).
26. treatment with monoamine oxidase inhibitors inhibitors or tricyclic antidepressants.
27. participation in another study.
28. more than eight puffs of salbutamol/day during the run-in period

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (42):
- Austria (6):
  - 205.334.4309 Boehringer Ingelheim Investigational Site, Gänserndorf
  - 205.334.4308 Boehringer Ingelheim Investigational Site, Hallein
  - 205.334.4306 Boehringer Ingelheim Investigational Site, Leoben
  - 205.334.4301 Boehringer Ingelheim Investigational Site, Linz
  - 205.334.4302 Boehringer Ingelheim Investigational Site, Neumarkt am Wallersee
  - 205.334.4305 Boehringer Ingelheim Investigational Site, Salzburg
- Canada (9):
  - 205.334.1009 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 205.334.1003 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 205.334.1005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 205.334.1008 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 205.334.1004 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 205.334.1010 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 205.334.1001 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 205.334.1006 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 205.334.1007 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- France (9):
  - 205.334.3303A Boehringer Ingelheim Investigational Site, Beuvry
  - 205.334.3303B Boehringer Ingelheim Investigational Site, Beuvry
  - 205.334.3305A Boehringer Ingelheim Investigational Site, Créteil
  - 205.334.3301A Boehringer Ingelheim Investigational Site, Grenoble
  - 205.334.3304A Boehringer Ingelheim Investigational Site, Saint-Priest-en-Jarez
  - 205.334.3306A Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.334.3306B Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.334.3302A Boehringer Ingelheim Investigational Site, Toulouse
  - 205.334.3302B Boehringer Ingelheim Investigational Site, Toulouse
- Germany (6):
  - 205.334.4908 Boehringer Ingelheim Investigational Site, Berlin
  - 205.334.4909 Boehringer Ingelheim Investigational Site, Berlin
  - 205.334.4902 Boehringer Ingelheim Investigational Site, Cologne
  - 205.334.4904 Boehringer Ingelheim Investigational Site, Donaustauf
  - 205.334.4901 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 205.334.4907 Boehringer Ingelheim Investigational Site, Kiel
- Italy (6):
  - 205.334.39007 Boehringer Ingelheim Investigational Site, Catania
  - 205.334.39002 Boehringer Ingelheim Investigational Site, Gaiato Pavullo (mo)
  - 205.334.39004 Boehringer Ingelheim Investigational Site, Milan
  - 205.334.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 205.334.39005 Boehringer Ingelheim Investigational Site, Roma
  - 205.334.39006 Boehringer Ingelheim Investigational Site, Roma
- Russia (3):
  - 205.334.7001 Boehringer Ingelheim Investigational Site, Moscow
  - 205.334.7002 Boehringer Ingelheim Investigational Site, Moscow
  - 205.334.7003 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Sweden (3):
  - 205.334.46003 Boehringer Ingelheim Investigational Site, Jönköping
  - 205.334.46002 Boehringer Ingelheim Investigational Site, Lund
  - 205.334.46001 Boehringer Ingelheim Investigational Site, Uppsala

REFERENCES:
- [Derived] Magnussen H, Paggiaro P, Schmidt H, Kesten S, Metzdorf N, Maltais F. Effect of combination treatment on lung volumes and exercise endurance time in COPD. Respir Med. 2012 Oct;106(10):1413-20. doi: 10.1016/j.rmed.2012.05.011. Epub 2012 Jun 28. PMID 22749044
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/205/205.334_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participant flow data are presented by treatment sequence
Groups:
- Tiotropium + Salmeterol / Fluticasone + Salmeterol: Tio 18mcg o.d. + Sal 50mcg b.i.d. / Flu+Sal 500+50mcg b.i.d.
- Fluticasone + Salmeterol / Tiotropium + Salmeterol: Flu+Sal 500+50mcg b.i.d. / Tio 18mcg o.d. + Sal 50mcg b.i.d.
Period: Overall Study
Arm/Group | Tiotropium + Salmeterol / Fluticasone + Salmeterol | Fluticasone + Salmeterol / Tiotropium + Salmeterol
Started | 172 | 172
Completed | 149 | 151
Not Completed | 23 | 21
Not completed — Adverse Event | 10 | 6
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Individual different reasons | 4 | 3
Period: Period 1
Arm/Group | Tiotropium + Salmeterol / Fluticasone + Salmeterol | Fluticasone + Salmeterol / Tiotropium + Salmeterol
Started | 172 | 172
Completed | 158 | 161
Not Completed | 14 | 11
Not completed — Adverse Event | 7 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Individual different reasons | 2 | 3
Period: Period 2
Arm/Group | Tiotropium + Salmeterol / Fluticasone + Salmeterol | Fluticasone + Salmeterol / Tiotropium + Salmeterol
Started | 157 | 160
Completed | 149 | 151
Not Completed | 8 | 9
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Individual different reasons | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium + Salmeterol / Fluticasone + Salmeterol | Fluticasone + Salmeterol / Tiotropium + Salmeterol | Total
Number analyzed (Participants) | 172 | 172 | 344
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (7.5) | 60.6 (7.6) | 61.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 124 | 123 | 247

OUTCOME MEASURES:

1. Primary Outcome: Post-dose TGV(FRC) (After 8 Weeks)
Description: Post-dose TGV(FRC) (Thoracic Gas Volume; co-primary endpoint) after 8 weeks
Time Frame: 8 weeks
Population: FAS using imputed values. The full analysis set (FAS) was defined to include all treated patients with any post-dosing efficacy data after at least 4 weeks for both investigational treatments in TGV(FRC) or endurance time.
Measure: Mean (Standard Error); unit: Litres
Groups:
- Tiotropium + Salmeterol: Tio 18mcg o.d. + Sal 50mcg b.i.d. in Period 1 or 2
- Fluticasone + Salmeterol: Flu+Sal 500+50mcg b.i.d. in Period 1 or 2
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 4.99 (0.07) | 5.07 (0.07)
Statistical Analysis 1: Comparison: Tiotropium + Salmeterol vs Fluticasone + Salmeterol; Test type: Superiority or Other; p = 0.0482, ANOVA; ANOVA with fixed terms for sequence, treatment, and period and random term for subject within sequence; Mean Difference (Final Values) = -0.087, 95% CI 2-sided [-0.174 to -0.001], Standard Error of Mean 0.044

2. Primary Outcome: Endurance Time (After 8 Weeks)
Description: Endurance time to the point of symptom limitation after 8 weeks during a constant work rate exercise test at 75% Wcap (co-primary endpoint)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Seconds | 463 (375) [316 to 691] | 453 (413) [307 to 720]
Statistical Analysis 1: Comparison: Tiotropium + Salmeterol vs Fluticasone + Salmeterol; Test type: Superiority or Other; p = 0.3407, Wilcoxon signed-rank test; Median Difference (Final Values) = 3.0, 95% CI 2-sided [-9.5 to 27.5] — The confidence interval was determined by Hodges-Lehmann method

3. Secondary Outcome: Post-dose TGV(FRC) (After 4 Weeks)
Description: Post-dose TGV(FRC) (Thoracic Gas Volume) after 4 weeks
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Litres | 5.00 (0.07) | 5.19 (0.07)

4. Secondary Outcome: Endurance Time (After 4 Weeks)
Description: Endurance time to the point of symptom limitation after 4 weeks during a constant work rate exercise test at 75% Wcap (co-primary endpoint)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Seconds | 458 (331) [343 to 674] | 450 (375) [301 to 676]

5. Secondary Outcome: Static Lung Volumes
Description: Trough TGV(FRC) (Thoracic Gas Volume) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 5.24 (0.08) | 5.25 (0.08)

6. Secondary Outcome: Static Lung Volumes
Description: Trough TGV(FRC) (Thoracic Gas Volume) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 5.32 (0.08) | 5.34 (0.08)

7. Secondary Outcome: Static Lung Volumes
Description: Trough RV (Residual Volume) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 4.23 (0.08) | 4.25 (0.08)

8. Secondary Outcome: Static Lung Volumes
Description: Trough RV (Residual Volume) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Litres | 4.28 (0.08) | 4.35 (0.08)

9. Secondary Outcome: Static Lung Volumes
Description: Post-dose RV (Residual Volume) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 3.92 (0.07) | 4.07 (0.07)

10. Secondary Outcome: Static Lung Volumes
Description: Post-dose RV (Residual Volume) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Litres | 3.91 (0.07) | 4.14 (0.07)

11. Secondary Outcome: Static Lung Volumes
Description: Trough IC (Inspiratory Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 2.33 (0.04) | 2.23 (0.04)

12. Secondary Outcome: Static Lung Volumes
Description: Trough IC (Inspiratory Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Litres | 2.28 (0.04) | 2.23 (0.04)

13. Secondary Outcome: Static Lung Volumes
Description: Post-dose IC (Inspiratory Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 2.47 (0.04) | 2.35 (0.04)

14. Secondary Outcome: Static Lung Volumes
Description: Post-dose IC (Inspiratory Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Litres | 2.46 (0.05) | 2.37 (0.05)

15. Secondary Outcome: Static Lung Volumes
Description: Trough IRV (Inspiratory Reserve Volume) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 280 | 281
Litres | 1.48 (0.04) | 1.41 (0.04)

16. Secondary Outcome: Static Lung Volumes
Description: Trough IRV (Inspiratory Reserve Volume) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 280 | 280
Litres | 1.47 (0.04) | 1.42 (0.04)

17. Secondary Outcome: Static Lung Volumes
Description: Post-dose IRV (Inspiratory Reserve Volume) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 280 | 281
Litres | 1.62 (0.04) | 1.55 (0.04)

18. Secondary Outcome: Static Lung Volumes
Description: Post-dose IRV (Inspiratory Reserve Volume) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 280 | 280
Litres | 1.62 (0.04) | 1.55 (0.04)

19. Secondary Outcome: Static Lung Volumes
Description: Trough TLC (Total Lung Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 7.47 (0.09) | 7.39 (0.09)

20. Secondary Outcome: Static Lung Volumes
Description: Trough TLC (Total Lung Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Litres | 7.52 (0.09) | 7.51 (0.09)

21. Secondary Outcome: Static Lung Volumes
Description: Post-dose TLC (Total Lung Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 7.36 (0.09) | 7.36 (0.09)

22. Secondary Outcome: Static Lung Volumes
Description: Post-dose TLC (Total Lung Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Litres | 7.33 (0.09) | 7.47 (0.09)

23. Secondary Outcome: Static Lung Volumes (Percent)
Description: Trough RV/TLC (Residual Volume over Total Lung Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of RV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of RV over TLC | 56.10 (0.54) | 57.18 (0.54)

24. Secondary Outcome: Static Lung Volumes (Percent)
Description: Trough RV/TLC (Residual Volume over Total Lung Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of RV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Percent of RV over TLC | 56.57 (0.56) | 57.47 (0.56)

25. Secondary Outcome: Static Lung Volumes (Percent)
Description: Post-dose RV/TLC (Residual Volume over Total Lung Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of RV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of RV over TLC | 52.79 (0.54) | 55.02 (0.54)

26. Secondary Outcome: Static Lung Volumes (Percent)
Description: Post-dose RV/TLC (Residual Volume over Total Lung Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of RV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Percent of RV over TLC | 53.09 (0.57) | 55.07 (0.57)

27. Secondary Outcome: Static Lung Volumes (Percent)
Description: Trough TGV/TLC (Thoracic Gas Volume over Total Lung Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of TGV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of TGV over TLC | 69.87 (0.47) | 70.94 (0.47)

28. Secondary Outcome: Static Lung Volumes (Percent)
Description: Trough TGV/TLC (Thoracic Gas Volume over Total Lung Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of TGV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Percent of TGV over TLC | 70.59 (0.47) | 70.99 (0.47)

29. Secondary Outcome: Static Lung Volumes (Percent)
Description: Post-dose TGV/TLC (Thoracic Gas Volume over Total Lung Capacity) after 8 weeks (measured by bodyphlethysmography)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of TGV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of TGV over TLC | 67.65 (0.49) | 68.85 (0.49)

30. Secondary Outcome: Static Lung Volumes (Percent)
Description: Post-dose TGV/TLC (Thoracic Gas Volume over Total Lung Capacity) after 4 weeks (measured by bodyphlethysmography)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of TGV over TLC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 307
Percent of TGV over TLC | 68.43 (0.49) | 69.22 (0.49)

31. Secondary Outcome: Slow Vital Capacity (SVC)
Description: Trough SVC (Slow Vital Capacity) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 306 | 304
Litres | 3.22 (0.05) | 3.12 (0.05)

32. Secondary Outcome: Slow Vital Capacity (SVC)
Description: Trough SVC (Slow Vital Capacity) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 305 | 301
Litres | 3.19 (0.05) | 3.12 (0.05)

33. Secondary Outcome: Slow Vital Capacity (SVC)
Description: Post-dose SVC (Slow Vital Capacity) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 306 | 304
Litres | 3.42 (0.05) | 3.28 (0.05)

34. Secondary Outcome: Slow Vital Capacity (SVC)
Description: Post-dose SVC (Slow Vital Capacity) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 305 | 301
Litres | 3.39 (0.05) | 3.27 (0.05)

35. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Trough FEV1 (Forced Expiratory Volume in 1 second) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 1.48 (0.03) | 1.44 (0.03)

36. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Trough FEV1 (Forced Expiratory Volume in 1 second) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Litres | 1.48 (0.03) | 1.45 (0.03)

37. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Post-dose FEV1 (Forced Expiratory Volume in 1 second) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 1.62 (0.03) | 1.55 (0.03)

38. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Post-dose FEV1 (Forced Expiratory Volume in 1 second) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Litres | 1.62 (0.03) | 1.55 (0.03)

39. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Trough percent predicted FEV1 (Forced Expiratory Volume in 1 second) according to ECCS after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of predicted FEV1
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of predicted FEV1 | 50.27 (0.78) | 49.12 (0.78)

40. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Trough percent predicted FEV1 (Forced Expiratory Volume in 1 second) according to ECCS after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of predicted FEV1
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Percent of predicted FEV1 | 50.40 (0.79) | 49.26 (0.79)

41. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Post-dose percent predicted FEV1 (Forced Expiratory Volume in 1 second) according to ECCS after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of predicted FEV1
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of predicted FEV1 | 54.99 (0.82) | 52.59 (0.82)

42. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Post-dose percent predicted FEV1 (Forced Expiratory Volume in 1 second) according to ECCS after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of predicted FEV1
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Percent of predicted FEV1 | 54.96 (0.82) | 52.64 (0.82)

43. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Trough FVC (Forced Vital Capacity) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 3.06 (0.05) | 2.94 (0.05)

44. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Trough FVC (Forced Vital Capacity) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Litres | 3.04 (0.05) | 2.93 (0.05)

45. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Post-dose FVC (Forced Vital Capacity) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Litres | 3.26 (0.05) | 3.11 (0.05)

46. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Post-dose FVC (Forced Vital Capacity) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Litres | 3.25 (0.05) | 3.11 (0.05)

47. Secondary Outcome: FEV1 Over FVC (Percent)
Description: Trough FEV1 (Forced Expiratory Volume in 1 second) over FVC (Forced Vital Capacity) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of FEV1 over FVC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of FEV1 over FVC | 49.16 (0.68) | 49.67 (0.68)

48. Secondary Outcome: FEV1 Over FVC (Percent)
Description: Trough FEV1 (Forced Expiratory Volume in 1 second) over FVC (Forced Vital Capacity) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of FEV1 over FVC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Percent of FEV1 over FVC | 49.74 (0.82) | 50.62 (0.82)

49. Secondary Outcome: FEV1 Over FVC (Percent)
Description: Post-dose FEV1 (Forced Expiratory Volume in 1 second) over FVC (Forced Vital Capacity) after 8 weeks (measured by spirometry)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of FEV1 over FVC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Percent of FEV1 over FVC | 50.77 (0.72) | 50.66 (0.72)

50. Secondary Outcome: FEV1 Over FVC (Percent)
Description: Post-dose FEV1 (Forced Expiratory Volume in 1 second) over FVC (Forced Vital Capacity) after 4 weeks (measured by spirometry)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Percent of FEV1 over FVC
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 308
Percent of FEV1 over FVC | 50.90 (0.73) | 50.91 (0.73)

51. Secondary Outcome: Symptom Intensity During Exercise
Description: Isotime Borg dyspnea scale after 8 weeks, Unit on a Scale (min. 0, max 10), 0 = no dyspnea, 10 = worst imaginable dyspnea
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Unit on a Scale
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Unit on a Scale | 4.77 (0.13) | 4.98 (0.13)

52. Secondary Outcome: Symptom Intensity During Exercise
Description: Isotime Borg dyspnea scale after 4 weeks, Unit on a Scale (min. 0, max. 10), 0 = no dyspnea, 10 = worst imaginable dyspnea
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Unit on a Scale
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Unit on a Scale | 4.80 (0.13) | 5.02 (0.13)

53. Secondary Outcome: Symptom Intensity During Exercise
Description: Isotime Borg leg discomfort scale after 8 weeks, Unit on a Scale (min. 0, max. 10), 0 = no leg dyscomfort, 10 = worst imaginable leg dyscomfort
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Unit on a Scale
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Unit on a Scale | 4.64 (0.15) | 4.53 (0.15)

54. Secondary Outcome: Symptom Intensity During Exercise
Description: Isotime Borg leg discomfort scale after 4 weeks, Unit on a Scale (min. 0, max. 10), 0 = no leg dyscomfort, 10 = worst imaginable leg dyscomfort
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Mean (Standard Error); unit: Unit on a Scale
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Unit on a Scale | 4.63 (0.15) | 4.63 (0.15)

55. Secondary Outcome: Dyspnea and Leg Discomfort
Description: Peak Borg dyspnea scale after 8 weeks, Unit on a Scale (min. 0, max 10)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Unit on a Scale | 6.52 (2.36) | 6.61 (2.31)

56. Secondary Outcome: Dyspnea and Leg Discomfort
Description: Peak Borg leg discomfort scale after 8 weeks, Unit on a Scale (min. 0, max 10)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Unit on a Scale | 6.10 (3.03) | 5.86 (3.01)

57. Secondary Outcome: Locus of Symptom Limitation at Peak Exercise During Exercise
Description: Reason for stopping exercise at baseline (leg discomfort, breathing discomfort, both or none)
Time Frame: baseline
Population: FAS using imputed values
Measure: Number; unit: Participants
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Participants
  Leg discomfort | 53 | 53
  Breathing discomfort | 132 | 132
  Both (leg and breathing discomfort) | 92 | 92
  None | 32 | 32

58. Secondary Outcome: Locus of Symptom Limitation at Peak Exercise During Exercise
Description: Reason for stopping exercise after 4 weeks (leg discomfort, breathing discomfort, both or none)
Time Frame: 4 weeks
Population: FAS using imputed values
Measure: Number; unit: Participants
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Participants
  Leg discomfort | 89 | 72
  Breathing discomfort | 104 | 119
  Both (leg and breathing discomfort) | 78 | 78
  None | 38 | 40

59. Secondary Outcome: Locus of Symptom Limitation at Peak Exercise During Exercise
Description: Reason for stopping exercise after 8 weeks (leg discomfort, breathing discomfort, both or none)
Time Frame: 8 weeks
Population: FAS using imputed values
Measure: Number; unit: Participants
Arm/Group | Tiotropium + Salmeterol | Fluticasone + Salmeterol
Number analyzed (Participants) | 309 | 309
Participants
  Leg discomfort | 88 | 72
  Breathing discomfort | 112 | 131
  Both (leg and breathing discomfort) | 82 | 78
  None | 27 | 28

ADVERSE EVENTS:
Time Frame: From drug administration until end of second treatment period plus 30 days.
Groups:
- Tiotropium + Salmeterol (Period 1): Tio 18mcg o.d. + Sal 50mcg b.i.d. in Period 1
- Tiotropium + Salmeterol (Period 2): Tio 18mcg o.d. + Sal 50mcg b.i.d. in Period 2
- Fluticasone + Salmeterol (Period 1): Flu+Sal 500+50mcg b.i.d. in Period 1
- Fluticasone + Salmeterol (Period 2): Flu+Sal 500+50mcg b.i.d. in Period 2
Arm/Group | Tiotropium + Salmeterol (Period 1) | Tiotropium + Salmeterol (Period 2) | Fluticasone + Salmeterol (Period 1) | Fluticasone + Salmeterol (Period 2)
Serious Adverse Events (participants affected / at risk) | 7/172 | 5/160 | 4/172 | 4/157
Other Adverse Events (participants affected / at risk) | 18/172 | 18/160 | 21/172 | 12/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium + Salmeterol (Period 1) (N=172) | Tiotropium + Salmeterol (Period 2) (N=160) | Fluticasone + Salmeterol (Period 1) (N=172) | Fluticasone + Salmeterol (Period 2) (N=157)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 2
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Musculeskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium + Salmeterol (Period 1) (N=172) | Tiotropium + Salmeterol (Period 2) (N=160) | Fluticasone + Salmeterol (Period 1) (N=172) | Fluticasone + Salmeterol (Period 2) (N=157)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 11 | 12 | 7
Nasopharyngitis (Infections and infestations) | 3 | 9 | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.